CLINICAL TRIAL: NCT01057667
Title: A Randomized, Double-blinded, Multicenter Study to Evaluate the Antiviral Efficacy and Safety of Adding the HCV Polymerase Inhibitor Prodrug (RO5024048) for 24 Weeks to the Currently Approved Combination of Pegasys® and Copegus® in Treatment-Naïve Patients With Chronic Hepatitis C Genotype 1 or 4
Brief Title: A Study of RO5024048 in Combination With Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin) in Patients With Chronic Hepatitis C Genotype 1 or 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV22621
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A: With RO5024048 (Experimental): Patients in arm A will receive RO5024048 (1000mg orally twice daily) for 24 weeks in addition to Pegasys (180 micrograms sc weekly) and Copegus (1000mg or 1200mg orally daily).
  Interventions: Drug: RO5024048; Drug: Ribavirin [Copegus]; Drug: peginterferon alfa-2a [Pegasys]
- Arm B: Standard treatment (Active Comparator): Patients in arm B will receive standard treatment with Pegasys (180 micrograms sc weekly) and Copegus (1000mg or 1200mg orally daily) for 48 weeks.
  Interventions: Drug: Ribavirin [Copegus]; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: RO5024048 — 1000mg bid po, 24 weeks
  Arms: Arm A: With RO5024048
Drug: Ribavirin [Copegus] — 1000mg or 1200mg po daily
Drug: peginterferon alfa-2a [Pegasys] — 180mcg sc weekly

SUMMARY:
This equally randomized (1:1), double-blind, parallel arm study will assess the safety and antiviral efficacy of RO5024048 added to standard Pegasys (peginterferon alfa-2a) plus Copegus (ribavirin) therapy in patients with chronic hepatitis C genotype 1 or 4. Patients in arm A will receive RO5024048 (1000mg orally twice daily) for 24 weeks in addition to Pegasys (180 micrograms sc weekly) and Copegus (1000mg or 1200mg orally daily). Patients achieving a rapid virological response (RVR) at week 4, sustained through week 22, will stop all treatment at week 24; non-RVR patients will continue treatment with Pegasys and Copegus for another 24 weeks up to week 48. Patients in arm B will receive standard treatment with Pegasys (180 micrograms sc weekly) and Copegus (1000mg or 1200mg orally daily) for 48 weeks. Anticipated time on study treatment is up to 48 weeks. Target sample size is <200.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age
* hepatitis C, genotype 1 or 4, of over 6 months duration
* treatment-naïve
* negative pregnancy test; female patients of childbearing age and male patients with female partners of childbearing age must use two forms of contraception during treatment and following the last dose of ribavirin in accordance with locally approved label for ribavirin

Exclusion Criteria:

* pregnant or breast feeding females or male partners of pregnant females
* previous interferon or ribavirin based therapy or investigational anti-HCV agent
* systemic antiviral therapy with established or perceived activity against HCV </=3 months prior to first dose of study drug
* hepatitis A or B, or HIV infection
* history or evidence of medical condition associated with chronic liver disease other than HCV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (undetectable HCV DNA as measured by Roche COBAS TaqMan HCV test) | 24 weeks after last treatment dose

SECONDARY OUTCOMES:
Virologic response over time | weeks 4, 12, 24, 36, 48 and 60
Pharmacokinetics of RO4995855 when RO5024048 is administered with peginterferon alfa-2a and ribavirin | week 12 and 24
Resistance profile of RO5024048 | weeks 1-24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (17):
  - La Jolla, California
  - Bradenton, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Albuquerque, New Mexico
  - New York, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Ottawa, Ontario

REFERENCES:
- [Derived] Tong X, Le Pogam S, Li L, Haines K, Piso K, Baronas V, Yan JM, So SS, Klumpp K, Najera I. In vivo emergence of a novel mutant L159F/L320F in the NS5B polymerase confers low-level resistance to the HCV polymerase inhibitors mericitabine and sofosbuvir. J Infect Dis. 2014 Mar 1;209(5):668-75. doi: 10.1093/infdis/jit562. Epub 2013 Oct 23. PMID 24154738